CLINICAL TRIAL: NCT05522634
Title: The Efficacy and Safety of Chinese Herbal Compound TJAOA101 in the Treatment of POI: A Multicenter, Prospective and Before-after Study.
Brief Title: A Clinical Study of Chinese Herbal Compound TJAOA101 in the Treatment of Premature Ovarian Insufficiency
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Shixuan Wang, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20220634-POI
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Premature Ovarian Failure
Keywords: Premature Ovarian Failure; Traditional Chinese Medicine
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TJAOA101 (Experimental): Once enrolled, participants will be administrated TJAOA101 and followed by a 3-month medication cycle. The usage of this herbal compound is to take orally twice a day(two sacks per). Add it to about 200ml warm water and take it half an hour before breakfast in the morning and half an hour before bedtime in the evening except menstrual period.
  Interventions: Drug: TJAOA101

INTERVENTIONS:
Drug: TJAOA101 — Once enrolled, participants will be administrated TJAOA101

SUMMARY:
Premature ovarian insufficiency (POI) seriously affects the physical and mental health of women. Nowadays, Chinese herbs have huge appeal and potential in treating POI. We have created a new Chinese herbal combination TJAOA101, whereas its safety and efficacy still need to be validated. Hence, we will perform a population-based, multicenter study to confirm the safety and efficacy of TJAOA101 in therapy of POI. We aim to provide a solid evidence for TCM in therapy of POI.

DETAILED DESCRIPTION:
Premature ovarian insufficiency (POI) seriously affects the physical and mental health of women. Nowadays, Chinese herbs have huge appeal and potential in treating POI. We have created a new Chinese herbal combination TJAOA101, whereas its safety and efficacy still need to be validated in multi-center and prospective clinical trials. We are conducting a prospective and before-after clinic trial with 100 eligible women aged 18-40 diagnosed POI will be participated. All participants will be administrated TJAOA101 drug twice every day for overall 3 months. The primary outcomes will be the basal level of serum FSH. The second outcome is the recovery rate of menstruation. All the outcomes will be assessed at baseline and 1, 2, 3 months following the 3 months' treatment. Adverse events(AEs) of patients will be assessed during the follow-up. The study was approved by the Medical Ethics Committee of the Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology (TJ-IRB20220634) according to the submitted study protocol (V.2.1, 10 May 2022) and informed consent (V.2.1, 10 May 2022). The results will be presented at domestic and international conferences and published in peer reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

1. The age range of patient is 18-40 years old.
2. The diagnostic criteria for POI is as follows: Age <40; and menopause or sporadic menstruation for more than 4 months; and bFSH>25 mIU/ml (the interval between two reexaminations should be more than one month, both reached this level)
3. Sign the informed consent form.

Exclusion Criteria:

1. Patient is known to be allergic or unsuitable for the Chinese herbal compound.
2. Women who are pregnant and lactating.
3. Patients had been menopause for more than 1 year.
4. Abnormal uterine bleeding, except ovulation disorders.
5. Women is taking hormone drugs and has stopped taking them within 3 months;
6. Women with endometriosis, myadenosis, submucosal fibroids or the size of non- submucosal fibroids is more than 4 cm.
7. The nature of pelvic mass is unknown.
8. Women with polycystic ovary syndrome, hyperprolactinemia, hyperandrogenemia, diabetes, thyroid and adrenal dysfunction and other endocrine diseases affecting ovulation.
9. Patients with serious primary diseases such as cardiovascular, liver, kidney, lung, biliary, hematopoietic system (Hb<90g/L) and malignant tumor, and psychiatric patients.
10. Patients are participating in other clinical trials or have participated in other clinical trials within the last month.
11. Unsuitable for the study evaluated by the investigator.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
recovery rate of ovarian function | 6 months
  As the definition of POI is based on menstruation and bFSH, the recovery of ovarian function is also based on the recovery of these indicators. In this study, the recovery of ovarian function is defined as serum bFSH decreased more than 50%, or recover to normal level; or two consecutive periods return to normal.

SECONDARY OUTCOMES:
serum AMH | 6 months
  serum AMH increased more than 50%, or recover to normal level.

CONTACTS AND LOCATIONS:
Overall Officials: Shixuan Wang, Professor, Study Chair — Department of Obstetrics and Gynecology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China